CLINICAL TRIAL: NCT01770093
Title: Preferences of Parents for Pediatric Inpatient Ward Physicians' Attire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0094-23-HYMC
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Parents; Physicians
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Parents of Pediatric Inpatients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
Several studies have been conducted throughout the world to evaluate patients' and parents' preferences regarding physicians' attire. Most studies have shown that the attire influences their feelings trust and confidence regarding their care. In most countries the preference is for formal attire. In other places a more casual attire is generally accepted. Israel is a country where casual dress is acceptable in most settings. Israeli physician's dress code has been discussed in the past, but has never been systematically studied. The aim of this study is to systematically examine the attitudes of parents of children who have been admitted to the pediatric ward towards physicians' attire.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose children have been hospitalized

Exclusion Criteria:

* All others

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents whose children have been hospitalized
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of parents preferring formal physician attire | Three years
  Final analysis of survey will be processed and the total number of parents preferring formal physician attire will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel